CLINICAL TRIAL: NCT01257607
Title: A Phase 2, Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of 1% MIM-D3 and 5% MIM-D3 Ophthalmic Solutions in the Environment, and During Challenge in the Controlled Adverse Environmental (CAE) Model
Brief Title: Safety and Efficacy Study of MIM-D3 Ophthalmic Solution for the Treatment of Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mimetogen Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIM-724
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1% MIM-D3 Ophthalmic Solution (Experimental)
  Interventions: Drug: MIM-D3 Ophthalmic Solution
- 5% MIM-D3 Ophthalmic Solution (Experimental)
  Interventions: Drug: MIM-D3 Ophthalmic Solution
- Placebo Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: MIM-D3 Ophthalmic Solution — 28 Days, BID
  Arms: 1% MIM-D3 Ophthalmic Solution; 5% MIM-D3 Ophthalmic Solution
Drug: Placebo Ophthalmic Solution — 28 Days, BID
  Arms: Placebo Ophthalmic Solution

SUMMARY:
The objective of this study is to compare the safety and efficacy of 1% MIM-D3 and 5% MIM-D3 to placebo for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age
2. Provide written informed consent
3. Have a reported history of dry eye
4. Have a history of use or desire to use eye drops for dry eye

Exclusion Criteria:

1. Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation (e.g. follicular conjunctivitis) at Visit 1, or have been diagnosed with ocular rosacea, or any viral or bacterial disease of the cornea or conjunctiva, within the last 12 months
2. Have any planned ocular and/or lid surgeries over the study period
3. Have corrected visual acuity greater than or equal to +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at Visit 1
4. Have an uncontrolled systemic disease
5. Be a woman who is pregnant, nursing or planning a pregnancy
6. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study
7. Have a known allergy and/or sensitivity to the test article or its components
8. Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
9. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 45 days of Visit 1
10. Be unable or unwilling to follow instructions, including participation in all study assessments and visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Corneal staining | 28 days
  Ocular surface damage

SECONDARY OUTCOMES:
Tear film break-up time | 42 days
Conjunctival redness | 42 days
Tear osmolarity | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates; John Lonsdale, MD, Principal Investigator — Central Maine Eye Care
Locations (1):
- Ora, Inc., Andover, Massachusetts, United States